CLINICAL TRIAL: NCT00458835
Title: A Randomized, Open-label, Single-dose, 3-period Crossover, Pharmacokinetic Study Designed to Compare the Systemic Des-ciclesonide Exposure of OMNARIS™ (Ciclesonide) Nasal Spray, Ciclesonide HFA Nasal Aerosol, and Orally Inhaled Ciclesonide
Brief Title: Comparison Between Systemic Exposure to Ciclesonide Nasal Spray, Ciclesonide HFA Nasal Aerosol and Orally Inhaled Ciclesonide (BY9010/M1-422)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Covis Pharma S.à.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BY9010/M1-422
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — ciclesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ciclesonide 300 mcg intranasally via aqueous nasal spray (Active Comparator)
  Interventions: Drug: Ciclesonide
- Ciclesonide 300 mcg intranasally via HFA nasal aerosol (Active Comparator)
  Interventions: Drug: Ciclesonide
- Ciclesonide 320 mcg orally inhaled via HFA MDI (Active Comparator)
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The purpose of this study is to compare the systemic des-ciclesonide exposure of OMNARIS™ (ciclesonide) nasal spray, ciclesonide HFA nasal aerosol, and orally inhaled ciclesonide HFA-metered-dose inhaler (MDI). The administration of the study medication will be as follows: three single doses, separated by a wash-out period. The study will provide further data on the safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent and HIPAA
* Body weight as indicate by a Body Mass Index (BMI) between ≥ 18 and ≤ 28 kg/m², and a body weight >50 kg
* General good health
* Ability to use oral inhaler

Main Exclusion Criteria:

* Pregnancy, breast feeding, intention to become pregnant during the course of the study or lack of safe contraception in pre-menopausal women
* Participation in any investigational drug trial within the 30 days before Screening Visit and thereafter
* History or current clinically relevant allergies or idiosyncrasy to drugs or food
* History of allergic reactions to any corticosteroids including ciclesonide or any excipients of the formulations
* Any contraindication to nasally administered corticosteroids
* History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, acute or chronic sinusitis, flu, severe acute respiratory syndrome (SARS)] within the 30 days before Screening Visit, or development of a respiratory infection during the Screening Period
* History or current evidence of any other relevant allergic, cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, metabolic, neurological, psychiatric, or other disease within the last 2 years
* Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding Screening Visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- ALTANA Pharma, Austin, Texas, United States

REFERENCES:
- [Derived] Nave R, Herzog R, Laurent A, Wingertzahn MA. Pharmacokinetics of ciclesonide and desisobutyryl ciclesonide after administration via aqueous nasal spray or hydrofluoroalkane nasal aerosol compared with orally inhaled ciclesonide: an open-label, single-dose, three-period crossover study in healthy volunteers. Clin Ther. 2009 Dec;31(12):2988-99. doi: 10.1016/j.clinthera.2009.12.002. PMID 20110036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 3-period crossover study of 30 subjects total; There were three single dose treatment periods separated by a washout of 7-14 days.
Groups:
- Ciclesonide Nasal Spray, Then Ciclesonide Nasal Aerosol, Then Ciclesonide HFA MDI: Participants first received Ciclesonide 300 mcg intranasally via aqueous nasal spray. After a 7-14 days washout period, they then received Ciclesonide 300 mcg via HFA nasal aerosol. After another 7-14 days washout period, they then received Ciclesonide 320 mcg orally inhaled via HFA MDI.
- Ciclesonide Nasal Aerosol, Then Ciclesonide HFA MDI, Then Ciclesonide Nasal Spray: Participants first received Ciclesonide 300 mcg via HFA nasal aerosol. After a 7-14 days washout period, they then received Ciclesonide 320 mcg orally inhaled via HFA MDI. After another 7-14 days washout period, they then received Ciclesonide 300 mcg intranasally via aqueous nasal spray.
- Ciclesonide HFA MDI, Then Ciclesonide Nasal Spray, Then Ciclesonide Nasal Aerosol: Participants first received Ciclesonide 320 mcg orally inhaled via HFA MDI. After a 7-14 days washout period, they then received Ciclesonide 300 mcg intranasally via aqueous nasal spray. After another 7-14 days washout period, they then received Ciclesonide 300 mcg via HFA nasal aerosol.
- Ciclesonide Nasal Spray, Then Ciclesonide HFA MDI, Then Ciclesonide Nasal Aerosol: Participants first received Ciclesonide 300 mcg intranasally via aqueous nasal spray. After a 7-14 days washout period, they then received Ciclesonide 320 mcg orally inhaled via HFA MDI. After another 7-14 days washout period, they then received Ciclesonide 300 mcg via HFA nasal aerosol.
- Ciclesonide Nasal Aerosol, Then Ciclesonide Nasal Spray, Then Ciclesonide HFA MDI: Participants first received Ciclesonide 300 mcg via HFA nasal aerosol. After a 7-14 days washout period, they then received Ciclesonide 300 mcg intranasally via aqueous nasal spray. After another 7-14 days washout period, they then received Ciclesonide 320 mcg orally inhaled via HFA MDI.
- Ciclesonide HFA MDI, Then Ciclesonide Nasal Aerosol, Then Ciclesonide Nasal Spray: Participants first received Ciclesonide 320 mcg orally inhaled via HFA MDI. After a 7-14 days washout period, they then received they then received Ciclesonide 300 mcg via HFA nasal aerosol. After another 7-14 days washout period, Ciclesonide 300 mcg intranasally via aqueous nasal spray.
Period: Overall Study
Arm/Group | Ciclesonide Nasal Spray, Then Ciclesonide Nasal Aerosol, Then Ciclesonide HFA MDI | Ciclesonide Nasal Aerosol, Then Ciclesonide HFA MDI, Then Ciclesonide Nasal Spray | Ciclesonide HFA MDI, Then Ciclesonide Nasal Spray, Then Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray, Then Ciclesonide HFA MDI, Then Ciclesonide Nasal Aerosol | Ciclesonide Nasal Aerosol, Then Ciclesonide Nasal Spray, Then Ciclesonide HFA MDI | Ciclesonide HFA MDI, Then Ciclesonide Nasal Aerosol, Then Ciclesonide Nasal Spray
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Comparability of treatment groups at baseline was not formally assessed. Any differences in the treatment groups at baseline were assumed to be at random.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide Nasal Spray, Then Ciclesonide Nasal Aerosol, Then Ciclesonide HFA MDI | Ciclesonide Nasal Aerosol, Then Ciclesonide HFA MDI, Then Ciclesonide Nasal Spray | Ciclesonide HFA MDI, Then Ciclesonide Nasal Spray, Then Ciclesonide Nasal Aerosol | Ciclesonide Nasal Spray, Then Ciclesonide HFA MDI, Then Ciclesonide Nasal Aerosol | Ciclesonide Nasal Aerosol, Then Ciclesonide Nasal Spray, Then Ciclesonide HFA MDI | Ciclesonide HFA MDI, Then Ciclesonide Nasal Aerosol, Then Ciclesonide Nasal Spray | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 5 | 5 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (13.39) | 38.4 (4.75) | 38.2 (13.39) | 26.8 (7.24) | 38 (14.09) | 33.8 (8.58) | 35.90 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 4 | 3 | 2 | 19
  Male | 2 | 1 | 2 | 1 | 2 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 5 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Systemic Exposure Measured by AUC, ng*hr/L, (Area Under the Serum Concentration) of Des-ciclesonide With Ciclesonide Nasal Spray, and Ciclesonide HFA Nasal Aerosol and Orally Inhaled Ciclesonide.
Description: The primary pharmacokinetics comparisons between treatments will be that of 300 mcg OMNARIS™ [ciclesonide] nasal spray and 300 mcg ciclesonide nasal HFA aerosol vs. 320 mcg orally inhaled ciclesonide as a reference. At prespecified timepoints, blood samples were obtained from subjects. It was anticipated that only a limited number of des-ciclesonide concentrations would exceed the lower limit of quantification (LLOQ) of 10 pg/mL for ciclesonide aqueous nasal spray. AUC for the aqueous nasal spray could not be determined due to the fact that there were too few analysis samples that produced values above the LLOQ.
Time Frame: 5min, 15min, 30min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 22h, 24h following drug administration.
Population: A total of 30 healthy volunteers were randomized in the study. Thirty were included in the ITT population; 29 subjects were included in the PP population. All 30 were included in the safety population. A subject was completely excluded from PP analyses as a major violation (common cold) and also due to the number of scheduled blood sample collections that could not be obtained subsequent to this subject's request for premature termination from the study.
Measure: Median (Full Range); unit: ng*hr/L
Groups:
- Ciclesonide Nasal Spray: Ciclesonide 300 mcg intranasally via aqueous nasal spray
- Ciclesonide Nasal Aerosol: Ciclesonide 300 mcg intranasally via HFA nasal aerosol
- Ciclesonide HFA MDI: Ciclesonide 320 mcg orally inhaled via HFA MDI
Arm/Group | Ciclesonide Nasal Spray | Ciclesonide Nasal Aerosol | Ciclesonide HFA MDI
Number analyzed (Participants) | 29 | 29 | 29
ng*hr/L | NA [NA to NA] — AUC could not be determined due to the fact that there were too few analysis samples that produced values above the LLOQ. | 403.7 [175.8 to 684.3] | 2762 [1603 to 4301]

2. Secondary Outcome: Comparison of Systemic Exposure Measured by Cmax, pg/mL, (Highest Concentration of Drug in the Blood) of Des-ciclesonide With Ciclesonide Nasal Spray, and Ciclesonide HFA Nasal Aerosol and Orally Inhaled Ciclesonide.
Description: The primary pharmacokinetics comparisons between treatments will be that of 300 mcg OMNARIS™ [ciclesonide] nasal spray and 300 mcg ciclesonide nasal HFA aerosol vs. 320 mcg orally inhaled ciclesonide as a reference. At prespecified timepoints, blood samples were obtained from subjects. The Cmax may be available only for a limited number of subjects. Thus the focus of statistical PK analysis will be on descriptive statistics. In particular, mean and median for Cmax will be calculated using data from subjects with Cmax above LLOQ (Lower Limit of Quantitation) and from all subjects with Cmax below LLOQ imputed by 0.
Time Frame: 5min, 15min, 30min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 22h, 24h following drug administration.
Population: as for outcome 1
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Ciclesonide Nasal Spray | Ciclesonide Nasal Aerosol | Ciclesonide HFA MDI
Number analyzed (Participants) | 29 | 29 | 29
pg/mL | 20.05 [13.40 to 26.70] | 59.0 [21.8 to 111.0] | 602.0 [332.0 to 1120]

ADVERSE EVENTS:
Time Frame: The study duration was about 4-6 weeks per subject consisting of: • Two screening visits, • A total of three Treatment Periods of 2 days each, • Two washout intervals of 7 (up to 14) days each, and • A Follow-up visit.
Arm/Group | Ciclesonide Nasal Spray | Ciclesonide Nasal Aerosol | Ciclesonide HFA MDI
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 4/29 | 9/29 | 3/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide Nasal Spray (N=29) | Ciclesonide Nasal Aerosol (N=29) | Ciclesonide HFA MDI (N=29)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Operation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No